CLINICAL TRIAL: NCT04303156
Title: An Open-Label, Single-Dose Study to Evaluate the Pharmacokinetics of Islatravir (MK-8591) in Subjects With Severe Renal Impairment
Brief Title: Pharmacokinetics of Islatravir in Participants With Severe Renal Impairment (MK-8591-026)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8591-026; 2020-000153-27 (EudraCT Number); MK-8591-026 (Other: Merck Protocol Number)
Record Dates: First submitted 2020-03-09; First posted 2020-03-10 (Actual); Results first posted 2021-10-28 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-09

CONDITIONS: Human Immunodeficiency Virus (HIV) Infection
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — islatravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Severe Renal Impairment (Experimental): Participants with severe renal impairment received a single oral dose of 60 mg MK-8591 (Islatravir) administered in capsule form.
  Interventions: Drug: Islatravir
- Healthy (Experimental): Healthy participants received a single oral dose of 60 mg Islatravir administered in capsule form.
  Interventions: Drug: Islatravir

INTERVENTIONS:
Drug: Islatravir — Single oral dose of 60 mg Islatravir administered in capsule form
  Other Names: MK-8591

SUMMARY:
This study will evaluate the general tolerability and pharmacokinetics (PK) of a single 60 mg dose of MK-8591 (Islatravir) in participants with severe renal insufficiency, compared to participants in good health.

ELIGIBILITY:
Inclusion Criteria:

Healthy participants must have the following:

* Is in good health
* Has a body mass index (BMI) ≥18.5 and ≤40 kg/m2.
* Female is not pregnant or breastfeeding, and is not one of the following: a woman of childbearing potential (WOCBP); if a WOCBP, is using an acceptable contraceptive method, or is abstinent from heterosexual intercourse as their preferred and usual lifestyle; a WOCBP must have a negative highly sensitive pregnancy test within 24 hours before the first dose of study intervention

Renally impaired participants must have the following:

* With the exception of renal impairment, is in generally good health
* Has a BMI ≥ 18.5 and ≤ 40 kg/m2
* Female is not pregnant or breastfeeding, and is not one of the following: a woman of childbearing potential (WOCBP); if a WOCBP, is using an acceptable contraceptive method, or is abstinent from heterosexual intercourse as their preferred and usual lifestyle; a WOCBP must have a negative highly sensitive pregnancy test within 24 hours before the first dose of study intervention

Exclusion Criteria:

Healthy participants must have the following:

* Has a history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases.
* Is mentally or legally incapacitated, has significant emotional problems
* Has known hypersensitivity to the active substance or any of the excipients of the study drug
* Has a history of significant multiple and/or severe allergies (e.g. food, drug, latex allergy), or has had an anaphylactic reaction or significant intolerability (i.e. systemic allergic reaction) to prescription or non-prescription drugs or food.
* Is positive for hepatitis B surface antigen, hepatitis C antibodies or HIV.
* Had major surgery, donated or lost 1 unit of blood (approximately 500 mL) within prior 4 weeks
* Is taking medications to treat chronic medical conditions and/or conditions associated with renal disease
* Has participated in another investigational study within prior 4 weeks

Other exclusions for healthy participants:

* Does not agree to follow the smoking restrictions
* Consumes greater than 1 glass for women, or 2 glasses for men of alcoholic beverages per day
* Consumes excessive amounts,of caffeinated beverages per day.
* Is a regular user of cannabis, any illicit drugs or has a history of drug (including alcohol) abuse within approximately prior 3 months.

Renally impaired participants must have the following:

* Has a history or presence of renal artery stenosis.
* Has had a renal transplant or nephrectomy.
* Has rapidly fluctuating renal function as determined by historical measurements.
* Has known hypersensitivity to the active substance or any of the excipients of the study drug.
* Has a history of cancer (malignancy).
* Has a history of significant multiple and/or severe allergies (e.g. food, drug, latex allergy), or has had an anaphylactic reaction or significant intolerability (i.e. systemic allergic reaction) to prescription or non-prescription drugs or food.
* Is positive for hepatitis B surface antigen, hepatitis C antibodies or human immunodeficiency virus (HIV).
* Had major surgery, donated or lost 1 unit of blood (approximately 500 mL) within 4 weeks prior to the prestudy (screening) visit.
* Is taking medications to treat chronic medical conditions and/or conditions associated with renal disease and has not been on a stable regimen for at least 1 month and/or is unable to withhold the use of the medication(s) within 4 hours prior to and 8 hours after administration of the study drug.
* Has participated in another investigational study within 4 weeks (or 5 half-lives, whichever is greater) prior to the prestudy (screening) visit.

Other exclusions for renally impaired participants

* Does not agree to follow the smoking restrictions.
* Consumes greater than 1 glass for women, or 2 glasses for men of alcoholic beverages per day.
* Consumes excessive amounts of caffeinated beverages per day.
* Is a regular user of cannabis, any illicit drugs or has a history of drug (including alcohol) abuse within approximately 3 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2020-10-19 (Actual); Study Completion 2020-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (2):
- Clinical Pharmacology of Miami ( Site 0001), Miami, Florida, United States
- Charite Research Organisation GmbH ( Site 0003), Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Matthews RP, Cao Y, Patel M, Weissler VL, Bhattacharyya A, De Lepeleire I, Last S, Rondon JC, Vargo R, Stoch SA, Iwamoto M. Safety and Pharmacokinetics of Islatravir in Individuals with Severe Renal Insufficiency. Antimicrob Agents Chemother. 2022 Dec 20;66(12):e0093122. doi: 10.1128/aac.00931-22. Epub 2022 Nov 8. PMID 36346229

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male and females with severe renal impairment between the ages of 18 and 75 years old (inclusive), and healthy matched controls were enrolled in this study.
Groups:
- Severe Renal Impairment: Participants with severe renal impairment received a single oral dose of 60 mg Islatravir administered in capsule form.
Period: Overall Study
Arm/Group | Severe Renal Impairment | Healthy
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Severe Renal Impairment | Healthy | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.7 (12.9) | 58.8 (5.5) | 58.3 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 3 | 3 | 6
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 6 | 5 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From Time 0 to Infinity (AUC0-inf) of Plasma Islatravir (ISL)
Description: Participants were treated with islatravir (ISL), and blood samples were collected from pre-dose up to 168 hours post-dose to determine the concentration of plasma ISL. The 95% confidence interval was derived from a fixed effects model performed on natural log-transformed values.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 168 hours post-dose
Population: Participants who comply with the protocol sufficiently to ensure that generated data will be likely to exhibit the effects of treatment, according to the underlying scientific model. Compliance covers such considerations as exposure to treatment, availability of measurements and absence of important protocol deviations.
Measure: Geometric Mean (95% Confidence Interval); unit: hr*μM
Arm/Group | Severe Renal Impairment | Healthy
Number analyzed (Participants) | 6 | 6
hr*μM | 14.4 [11.8 to 17.6] | 6.54 [4.77 to 8.98]
Statistical Analysis 1: Comparison: Severe Renal Impairment vs Healthy; Geometric mean ratio (GMR); Test type: Other; GMR = 2.20, 90% CI 2-sided [1.68 to 2.88] — Severe Renal Impairment / Healthy; GMR calculated using the mean square error referencing a t-distribution. Confidence limits exponentiated to obtain the 90% confidence interval

2. Primary Outcome: Area Under the Curve From Time 0 to Last Sampling Time (AUC0-last) of Plasma ISL
Description: Participants were treated with ISL, and blood samples were collected from pre-dose up to 168 hours post-dose to determine the concentration of plasma ISL. The 95% confidence interval was derived from a fixed effects model performed on natural log-transformed values.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 168 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: hr*μM
Arm/Group | Severe Renal Impairment | Healthy
Number analyzed (Participants) | 6 | 6
hr*μM | 11.0 [9.17 to 13.1] | 5.68 [4.06 to 7.94]
Statistical Analysis 1: Comparison: Severe Renal Impairment vs Healthy; GMR; Test type: Other; GMR = 1.93, 90% CI 2-sided [1.46 to 2.55] — Severe Renal Impairment / Healthy; [other analysis details as in outcome 1, analysis 1]

3. Primary Outcome: Maximum Concentration (Cmax) of Plasma ISL
Description: as for outcome 2
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 168 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μM
Arm/Group | Severe Renal Impairment | Healthy
Number analyzed (Participants) | 6 | 6
μM | 1.23 [1.06 to 1.42] | 1.19 [0.699 to 2.04]
Statistical Analysis 1: Comparison: Severe Renal Impairment vs Healthy; GMR; Test type: Other; GMR = 1.03, 90% CI 2-sided [0.67 to 1.57] — Severe Renal Impairment / Healthy; [other analysis details as in outcome 1, analysis 1]

4. Primary Outcome: Time of Maximum Concentration (Tmax) of Plasma ISL
Description: Participants were treated with ISL, and blood samples were collected from pre-dose up to 168 hours post-dose to determine the concentration of plasma ISL. The Tmax of plasma ISL was expressed as a median.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 168 hours post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | Severe Renal Impairment | Healthy
Number analyzed (Participants) | 6 | 6
Hours | 1.03 [1.00 to 2.00] | 0.75 [0.5 to 1.00]

5. Primary Outcome: Apparent Terminal Half-life (t1/2) of Plasma ISL
Description: Participants were treated with ISL, and blood samples were collected from pre-dose up to 168 hours post-dose to determine the concentration of plasma ISL. The Geometric Coefficient of Variation was expressed as a percent (%CV), and is calculated from the square root of corresponding estimated variance obtained for each population in fixed effect model multiplied by 100.
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 168 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Severe Renal Impairment | Healthy
Number analyzed (Participants) | 6 | 6
Hours | 127 (7.7) | 72.0 (15.5)

6. Primary Outcome: Apparent Clearance (CL/F) of Plasma ISL
Description: as for outcome 2
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 168 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: L/hr
Arm/Group | Severe Renal Impairment | Healthy
Number analyzed (Participants) | 6 | 6
L/hr | 14.2 [11.6 to 17.4] | 31.3 [22.8 to 42.9]
Statistical Analysis 1: Comparison: Severe Renal Impairment vs Healthy; GMR; Test type: Other; GMR = 0.46, 90% CI 2-sided [0.35 to 0.60] — Severe Renal Impairment / Healthy; [other analysis details as in outcome 1, analysis 1]

7. Primary Outcome: Apparent Volume of Distribution (Vz/F) of Plasma ISL
Description: as for outcome 2
Time Frame: Pre-dose, 0.25, 0.5, 1, 2, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 168 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Liters
Arm/Group | Severe Renal Impairment | Healthy
Number analyzed (Participants) | 6 | 6
Liters | 2610 [2170 to 3140] | 3250 [2100 to 5030]
Statistical Analysis 1: Comparison: Severe Renal Impairment vs Healthy; GMR; Test type: Other; GMR = 0.80, 90% CI 2-sided [0.56 to 1.14] — Severe Renal Impairment / Healthy; [other analysis details as in outcome 1, analysis 1]

8. Secondary Outcome: AUC0-inf of ISL Triphosphate (ISL-TP) in Peripheral Blood Mononuclear Cells (PBMC)
Description: Participants were treated with ISL, and peripheral blood samples were collected from pre-dose up to 168 hours post-dose to determine the concentration of ISL-TP in PBMCs. The 95% confidence interval was derived from a fixed effects model performed on natural log-transformed values.
Time Frame: Pre-dose, 4, 24, 48, 96, 168 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: hr*pmol/10^6 cells
Arm/Group | Severe Renal Impairment | Healthy
Number analyzed (Participants) | 6 | 6
hr*pmol/10^6 cells | 5810 [3890 to 8700] | 3920 [2830 to 5420]
Statistical Analysis 1: Comparison: Severe Renal Impairment vs Healthy; GMR; Test type: Other; GMR = 1.48, 90% CI 2-sided [1.03 to 2.14] — Severe Renal Impairment / Healthy; [other analysis details as in outcome 1, analysis 1]

9. Secondary Outcome: AUC0-last of ISL-TP in PBMC
Description: Participants were treated with ISL and peripheral blood samples were collected from pre-dose up to 168 hours post-dose to determine the concentration of ISL-TP in PBMCs. The 95% confidence interval was derived from a fixed effects model performed on natural log-transformed values.
Time Frame: Pre-dose, 4, 24, 48, 96, 168 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: hr*pmol/10^6 cells
Arm/Group | Severe Renal Impairment | Healthy
Number analyzed (Participants) | 6 | 6
hr*pmol/10^6 cells | 5200 [3670 to 7370] | 3780 [2720 to 5230]
Statistical Analysis 1: Comparison: Severe Renal Impairment vs Healthy; GMR; Test type: Other; GMR = 1.38, 90% CI 2-sided [0.98 to 1.93] — Severe Renal Impairment / Healthy; [other analysis details as in outcome 1, analysis 1]

10. Secondary Outcome: Cmax of ISL-TP in PBMC
Description: as for outcome 9
Time Frame: Pre-dose, 4, 24, 48, 96, 168 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: pmol/10^6 cells
Arm/Group | Severe Renal Impairment | Healthy
Number analyzed (Participants) | 6 | 6
pmol/10^6 cells | 20.3 [15.1 to 27.4] | 21.6 [13.7 to 34.1]
Statistical Analysis 1: Comparison: Severe Renal Impairment vs Healthy; GMR; Test type: Other; GMR = 0.94, 90% CI 2-sided [0.64 to 1.39] — Severe Renal Impairment / Healthy; [other analysis details as in outcome 1, analysis 1]

11. Secondary Outcome: Tmax of ISL-TP in PBMC
Description: Participants were treated with ISL and peripheral blood samples were collected from pre-dose up to 168 hours post-dose to determine the concentration of ISL-TP in PBMCs. The Tmax of ISL-TP was expressed as a median.
Time Frame: Pre-dose, 4, 24, 48, 96, 168 hours post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | Severe Renal Impairment | Healthy
Number analyzed (Participants) | 6 | 6
Hours | 36.00 [24.00 to 240.12] | 24.00 [4.00 to 239.78]

12. Secondary Outcome: Concentration at 24 Hours Post Dose (C24) of ISL-TP in PBMC
Description: Participants were treated with ISL and peripheral blood samples were collected at 24 hours post-dose to determine the concentration of ISL-TP in PBMCs. The 95% confidence interval was derived from a fixed effects model performed on natural log-transformed values.
Time Frame: 24 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: pmol/10^6 cells
Arm/Group | Severe Renal Impairment | Healthy
Number analyzed (Participants) | 6 | 6
pmol/10^6 cells | 18.4 [14.2 to 23.8] | 19.0 [12.9 to 28.2]
Statistical Analysis 1: Comparison: Severe Renal Impairment vs Healthy; GMR; Test type: Other; GMR = 0.97, 90% CI 2-sided [0.69 to 1.35] — Severe Renal Impairment / Healthy; [other analysis details as in outcome 1, analysis 1]

13. Secondary Outcome: Concentration at 168 Hours Post Dose (C168) of ISL-TP in PBMC
Description: Participants were treated with ISL and peripheral blood samples were collected at 168 hours post-dose to determine the concentration of ISL-TP in PBMCs. The 95% confidence interval was derived from a fixed effects model performed on natural log-transformed values.
Time Frame: 168 hours post-dose
Population: Participants who comply with the protocol sufficiently to ensure that generated data will be likely to exhibit the effects of treatment, according to the underlying scientific model. Compliance covers such considerations as exposure to treatment, availability of measurements and absence of important protocol deviations. One sample was missing for a Healthy participant.
Measure: Geometric Mean (95% Confidence Interval); unit: pmol/10^6 cells
Arm/Group | Severe Renal Impairment | Healthy
Number analyzed (Participants) | 6 | 5
pmol/10^6 cells | 8.06 [4.69 to 13.9] | 4.43 [0.938 to 20.9]
Statistical Analysis 1: Comparison: Severe Renal Impairment vs Healthy; GMR; Test type: Other; GMR = 1.82, 90% CI 2-sided [0.55 to 6.02] — Severe Renal Impairment / Healthy; [other analysis details as in outcome 1, analysis 1]

14. Secondary Outcome: Concentration at 672 Hours Post Dose (C672) of ISL-TP in PBMC
Description: Participants were treated with ISL and peripheral blood samples were collected at 672 hours post-dose to determine the concentration of ISL-TP in PBMCs. The 95% confidence interval was derived from a fixed effects model performed on natural log-transformed values.
Time Frame: 672 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: pmol/10^6 cells
Arm/Group | Severe Renal Impairment | Healthy
Number analyzed (Participants) | 6 | 6
pmol/10^6 cells | 1.96 [0.982 to 3.92] | 0.730 [0.489 to 1.09]
Statistical Analysis 1: Comparison: Severe Renal Impairment vs Healthy; GMR; Test type: Other; GMR = 2.69, 90% CI 2-sided [1.51 to 4.80] — Severe Renal Impairment / Healthy; [other analysis details as in outcome 1, analysis 1]

15. Secondary Outcome: T1/2 of ISL-TP in PBMC
Description: Participants were treated with ISL, and blood samples were collected from pre-dose up to 168 hours post-dose to determine the concentration of ISL-TP in PBMCs. The t1/2 of plasma ISL was expressed as a geometric mean. The Geometric Coefficient of Variation was expressed as a percent (%CV), and is calculated from the square root of corresponding estimated variance obtained for each population in fixed effect model multiplied by 100.
Time Frame: Pre-dose, 4, 24, 48, 96, 168 hours post-dose
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Severe Renal Impairment | Healthy
Number analyzed (Participants) | 6 | 6
Hours | 181 (48.4) | 131 (19.0)

16. Secondary Outcome: Percentage of Participants With an Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Time Frame: Up to Day 29
Population: All participants who received at least one dose of treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Severe Renal Impairment | Healthy
Number analyzed (Participants) | 6 | 6
Percentage of participants | 16.7 | 0.0

17. Secondary Outcome: Percentage of Participants Who Discontinued From the Study Due to an AE
Description: as for outcome 16
Time Frame: Up to Day 29
Population: All participants who received at least one dose of treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Severe Renal Impairment | Healthy
Number analyzed (Participants) | 6 | 6
Percentage of participants | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) from day of treatment (Day 1) up to day 29. All-cause mortality from day of randomization (Day 1) up to day 29.
Description: For AEs the population analyzed consisted of all participants who received at least one dose of treatment. For All-cause mortality the population analyzed consisted of all randomized participants.
Arm/Group | Severe Renal Impairment | Healthy
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 1/6 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Severe Renal Impairment (N=6) | Healthy (N=6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-24): https://cdn.clinicaltrials.gov/large-docs/56/NCT04303156/Prot_SAP_000.pdf